CLINICAL TRIAL: NCT04624191
Title: Clinical Impact of Home Oxygen Saturation Measurement in Patients With Interstitial Lung Disease: Quality of Live, Health Care Use, Score of Anxiety, Depression and Dyspnea and Physical Activity Level
Brief Title: Clinical Impact of HOME Oxygen SATURation Measurement (SATURHOME)
Acronym: SATURHOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Fondation IUCPQ (Other)
Responsible Party: Principal Investigator, Geneviève Dion, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-3417
Record Dates: First submitted 2020-09-18; First posted 2020-11-10 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Interstitial Lung Disease
Keywords: Saturometry at home; Quality of life; Heath care use; Physical activity level
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group participants will be asked to measure their oxygen saturation on a daily basis.
  Interventions: Other: Saturation at home
- Control Group (No Intervention): Usual Care

INTERVENTIONS:
Other: Saturation at home — Clinical benefit of taking saturation at home in interstitial lung disease
  Arms: Intervention Group

SUMMARY:
The use of saturometry at home is more and more widespread in patients suffering from interstitial pulmonary diseases (IPD), the patients seeing it as reassurance and a concrete way to follow the evolution of their disease. However, there are no studies evaluating the real clinical benefit of taking saturation at home in this population. In addition, clinical experience seems rather to demonstrate an increase in the anxiety level and the number of clinically unnecessary consultations related to the use of this measure.

The secondary objectives are to determine the impact of this measurement on: (1) the health care use (telephone calls, medical consultations and hospitalizations), (2) dyspnea score, (3) the anxiety and depression score (HADS score) and (4) the physical activity level. The exploratory objectives will be to determine if the measurement of saturation at home makes it possible to (1) predict the occurrence of acute exacerbations of fibrosis, (2) effectively predict the decline in respiratory function tests and (3) 1-year mortality. The investigator will also assess whether this measure makes it possible to screen patients with oxygen therapy needs at home. The investigator hypothesize that measuring oxygen saturation at home will lead to a significant deterioration in quality of life, an increase in the use of health care, a significant increase in the rate of anxiety and depression, dyspnea and a decrease in the physical activity level.

DETAILED DESCRIPTION:
Measurement tools

1. Quality of life: King's Brief Interstitial Lung Disease
2. Anxiety and depression score: HADS score
3. Dyspnea score : UCSD questionnaire
4. Physical activity level during 7 days: MoveMonitor by McRoberts
5. Home base saturation: Nonin Ny vantagr 9590
6. Disease evolution : complete lung function (plethymography, sprimoetry, DLCO), 6-minute walking test (following the ATS recommandation)

ELIGIBILITY:
Inclusion Criteria:

* Fibrosing interstitial lung disease
* Saturation below 90% during the 6-minute walk test
* Clinically stable

Exclusion Criteria:

* Oxygen dependent at rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life by questionnaire | 1 year
  Impact of home base saturometry on quality of life

SECONDARY OUTCOMES:
Health care use (phone calls, medical consultation) | 1 year
  Impact of home base saturometry on health car use as number and principal reason for : telephone calls, medical consultations and hospitalizations.
Dyspnea score | 1 year
  Impact of home base saturometry on dyspnea score with the University of California, San Diego Shortness of breath Questionnaire (UCSD) in a scale between 0 to 120 where 120 is the worst score.
Anxiety and depression score | 1 year
  Impact of home base saturometry on anxiety and depression score with the Hospital Anxiety and Depression Scale Questionnaire (HADs) in a scale between 0 to 42, where 42 is the worst score.
Physical activity level | 1 year
  Impact of home base saturometry on physical activity level measure by accelerometer (McRoberts) and define by steps number.
Energy expenditure | 1 year
  Impact of home base saturometry on energy expenditure (number of kilocalories burn by day), measure by accelerometer (McRoberts).

OTHER OUTCOMES:
Acute exacerbation | 1 year
  Impact of home base saturometry on predict the occurrence of acute exacerbations of fibrosis.
  Occurence: number of exacerbation of fibrosis during the year.
Pulmonary function decline | 1 year
  Impact of home base saturometry on predict the decline in respiratory function tests, principally the forced vital capacity.
Mortality | 1 year
  Impact of home base saturometry on 1-year mortality prediction

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Dion, MD, Principal Investigator — Institut universitaire de pneumologie et cardiologue de Québec - ULaval
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No